CLINICAL TRIAL: NCT00618722
Title: Phase 1-2, Multicenter, Randomized, Placebo-Controlled, Parallel-Group Study of the Safety and Efficacy of ATX-101 (Sodium Deoxycholate for Injection) for the Reduction of Subcutaneous Fat in the Submental Area
Brief Title: Phase 1-2 Study of Deoxycholic Acid Injection (ATX-101) for the Reduction of Submental Fat
Acronym: ATX-101
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATX-101-06-03; 2007-000146-13 (EudraCT Number)
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-06

CONDITIONS: Moderate or Severe Submental Fullness
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Deoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Deoxycholic Acid Injection 1 mg/cm² (Experimental): Participants received 0.5% deoxycholic acid administered in 0.2 mL injections, up to 4.8 mL (1 mg/cm²) per treatment session at intervals of approximately 1 month for up to a maximum of 4 treatments.
  Interventions: Drug: Deoxycholic Acid Injection
- Deoxycholic acid Injection 2 mg/cm² (Experimental): Participants received 1.0% deoxycholic acid administered in 0.2 mL injections, up to 4.8 mL (2 mg/cm²) per treatment session at intervals of approximately 1 month for up to a maximum of 4 treatments.
  Interventions: Drug: Deoxycholic Acid Injection
- Deoxycholic acid Injection 4 mg/cm² (Experimental): Participants received 2.0% deoxycholic acid administered in 0.2 mL injections, up to 4.8 mL (4 mg/cm²) per treatment session at intervals of approximately 1 month for up to a maximum of 4 treatments.
  Interventions: Drug: Deoxycholic Acid Injection
- Placebo (Placebo Comparator): Participants received placebo administered in 0.2 mL injections, up to 4.8 mL per treatment session at intervals of approximately 1 month for up to a maximum of 4 treatments.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deoxycholic Acid Injection
  Other Names: ATX-101
  Arms: Deoxycholic Acid Injection 1 mg/cm²; Deoxycholic acid Injection 2 mg/cm²; Deoxycholic acid Injection 4 mg/cm²
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the safety and potential efficacy of deoxycholic acid injection compared to placebo for the reduction of submental fat (fat below the chin).

DETAILED DESCRIPTION:
The trial included an initial cohort (3 participants in each arm) to evaluate safety followed by expansion to a second, larger cohort if adequate safety was determined in the initial cohort. Data from both cohorts was pooled for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Submental fat (SMF) that was considered undesirable by the subject and graded by the investigator as 2 or 3 using the SMF rating scale
* Good general health
* Signed informed consent

Exclusion Criteria:

* History of any treatment in the neck or chin area
* Loose skin or prominent platysmal bands in the neck or chin area
* Recent treatment with anticoagulants
* Presence of clinically significant health problems

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Beddingfield, MD. PhD, Study Director — Kythera Biopharmaceuticals, Inc.
Locations (6):
- Australia (3):
  - Investigational Site, Carina Heights
  - Investigational Site, Gold Coast
  - Investigational Site, Toorak
- Canada (2):
  - Investigational Site, Oakville, Ontario
  - Investigational Site, Niagara Falls
- Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Goodman GJ, Spelman LJ, Lowe N, Bowen B. Randomized, Placebo-Controlled Phase 1/2 Study to Determine the Appropriate ATX-101 Concentration for Reduction of Submental Fat. Dermatol Surg. 2021 Aug 1;47(8):1065-1070. doi: 10.1097/DSS.0000000000003092. PMID 34115682

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 study centers: 1 in the United Kingdom, 2 in Canada, and 3 in Australia.
Pre-assignment Details: Enrollment was conducted in 2 stages, an initial cohort in which preliminary safety and tolerability were evaluated and a second cohort (contingent cohort), which was enrolled after it had been determined that acceptable safety and tolerability were observed in the initial cohort. Participants from both cohorts were pooled for analysis.
Period: Overall Study
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Deoxycholic Acid Injection 4 mg/cm² | Placebo
Started | 21 | 20 | 22 | 22
Received Treatment | 20 | 20 | 22 | 22
Completed | 18 | 18 | 19 | 18
Not Completed | 3 | 2 | 3 | 4
Not completed — Refusal of Treatment | 0 | 0 | 1 | 0
Not completed — Patient Request | 1 | 1 | 1 | 1
Not completed — Inability to Complete Study Procedure | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 2
Not completed — Miscellaneous Reasons | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Deoxycholic Acid Injection 4 mg/cm² | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 22 | 22 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (9.71) | 45.5 (7.37) | 44.4 (6.95) | 48.0 (9.78) | 45.5 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 11 | 13 | 56
  Male | 4 | 4 | 11 | 9 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20 | 19 | 22 | 21 | 82
  Black | 0 | 0 | 0 | 0 | 0
  Hispanic | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Other | 0 | 1 | 0 | 0 | 1
Weight [Mean (Standard Deviation); unit: kg] | 77.56 (14.022) | 68.53 (12.472) | 79.28 (12.950) | 80.13 (11.083) | 76.53 (13.239)
Submental Fat (SMF) Rating [Number; unit: participants] — SMF Ratings:
  * 0 = Absent submental convexity: No localized submental fat evident;
  * 1 = Mild submental convexity: Minimal, localized submental fat;
  * 2 = Moderate submental convexity: Prominent, localized submental fat;
  * 3 = Severe submental convexity: Marked, localized submental fat;
  * 4 = Extreme submental convexity.
  participants
    2 | 13 | 12 | 13 | 13 | 51
    3 | 7 | 8 | 9 | 9 | 33
Fitzpatrick Skin Type [Number; unit: participants] — Fitzpatrick Skin Type is a numerical classification schema for human skin color and typical response to ultraviolet (UV) light:
  * Type I: Pale white skin, blue/hazel eyes, blond/red hair; Always burns, does not tan.
  * Type II: Fair skin, blue eyes; Burns easily, tans poorly.
  * Type III: Darker white skin; Tans after initial burn.
  * Type IV: Light brown skin; Burns minimally, tans easily.
  * Type V: Brown skin; Rarely burns, tans darkly easily.
  * Type VI: Dark brown or black skin; Never burns, always tans darkly.
  participants
    I-III | 20 | 20 | 22 | 22 | 84
    IV-VI | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The investigator determined the relationship of each adverse event to the administration of study drug.
  Severity of adverse events was determined using the following scale:
  * Mild: The participant is aware of a sign or symptom, but it is easily tolerated
  * Moderate: Discomfort or interference with usual activity
  * Severe: Incapacitating, with inability to engage in usual activity.
  A serious AE (SAE) was defined as an event that may constitute a significant medical hazard or side-effect, regardless of the investigator or sponsor's opinion regarding relatedness to study material. Serious events included, but were not limited to, any event that:
  * was fatal
  * was life-threatening
  * required inpatient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * was a congenital anomaly/birth defect
  * other significant medical hazard
Time Frame: From the first dose of study drug until 12 weeks after the last dose (up to 24 weeks after first treatment).
Population: Safety and Modified Intent to Treat (mITT) population including all randomized participants who received at least 1 dose of study drug and who had at least 1 post-baseline observation.
Measure: Number; unit: participants
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Deoxycholic Acid Injection 4 mg/cm² | Placebo
Number analyzed (Participants) | 20 | 20 | 22 | 22
participants
  Any adverse event | 20 | 19 | 22 | 21
  Adverse event associated with treatment area | 20 | 19 | 21 | 20
  Study drug-related adverse event | 20 | 19 | 21 | 20
  Severe adverse event | 0 | 3 | 3 | 1
  Study drug-related severe adverse event | 0 | 1 | 2 | 0
  Serious adverse event | 0 | 0 | 0 | 0
  Discontinued due to adverse event | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Submental Fat (SMF) Rating Scale Score
Description: The SMF rating scale score is based on the investigator's clinical evaluation of the participant, where submental fullness is scored on a 5-point ordinal scale (0-4) with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme.
  A negative change from Baseline indicates improvement.
Time Frame: Baseline and 4 weeks after last treatment (up to 16 weeks after first dose)
Population: Safety/mITT population with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Deoxycholic Acid Injection 4 mg/cm² | Placebo
Number analyzed (Participants) | 17 | 19 | 19 | 20
units on a scale | -0.9 (0.70) | -0.8 (0.60) | -0.7 (0.75) | -0.5 (0.60)
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.043, ANCOVA; Based on analysis of covariance (ANCOVA) model with treatment as fixed effect and baseline SMF rating as covariate; LS Mean Difference = -0.4, 95% CI 2-sided [-0.9 to 0.0]
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.050, ANCOVA; Based on analysis of covariance (ANCOVA) model with treatment as fixed effect and baseline SMF rating as covariate; LS Mean Difference = -0.4, 95% CI 2-sided [-0.8 to 0.0]
Statistical Analysis 3: Comparison: Deoxycholic Acid Injection 4 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.249, ANCOVA; Based on analysis of covariance (ANCOVA) model with treatment as fixed effect and baseline SMF rating as covariate; LS Mean Difference = -0.2, 95% CI 2-sided [-0.7 to 0.2]

3. Secondary Outcome: Change From Baseline in Subject Satisfaction With Appearance Rating Scale
Description: The Subject Satisfaction with Appearance Rating Scale assesses participants' satisfaction with their appearance in association with the face and chin on a 7-point scale from 0 to 6 where 0 = Extremely dissatisfied, 1 = Dissatisfied, 2 = Slightly dissatisfied, 3 = Neither satisfied nor dissatisfied, 4 = Slightly satisfied, 5 = Satisfied and 6 = Extremely satisfied. A positive change from Baseline indicates improvement.
Time Frame: Baseline and 4 weeks after last treatment (up to 16 weeks after first dose)
Population: Safety/mITT population with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Deoxycholic Acid Injection 4 mg/cm² | Placebo
Number analyzed (Participants) | 17 | 18 | 18 | 20
units on a scale | 3.8 (1.85) | 3.3 (1.78) | 3.5 (1.42) | 1.9 (2.29)
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA; Based on analysis of covariance (ANCOVA) model with treatment as fixed effect and baseline SMF rating as covariate; LS Mean Difference = 1.9, 95% CI 2-sided [0.7 to 3.1]
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.030, ANCOVA; Based on analysis of covariance (ANCOVA) model with treatment as fixed effect and baseline SMF rating as covariate; LS Mean Difference = 1.4, 95% CI 2-sided [0.1 to 2.6]
Statistical Analysis 3: Comparison: Deoxycholic Acid Injection 4 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.012, ANCOVA; Based on analysis of covariance (ANCOVA) model with treatment as fixed effect and baseline SMF rating as covariate; LS Mean Difference = 1.6, 95% CI 2-sided [0.4 to 2.8]

4. Secondary Outcome: Percentage of Participants With a Response in the Subject Global Improvement Rating
Description: Participants were asked to rate their total improvement or worsening in the appearance and physical feeling of their chin and neck area since before they received study treatment, whether or not they believed it was due to study treatment or to any other cause.
  0 = Very much worse, 1 = Much worse, 2 = Minimally worse, 3 = No change, 4 = Minimally improved, 5 = Much improved, 6 = Very much improved.
  Response is defined as any improvement, ie, a global improvement rating of 4, 5, or 6.
Time Frame: 4 weeks after last treatment (up to 16 weeks after first dose)
Population: Safety/mITT population
Measure: Number; unit: percentage of participants
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Deoxycholic Acid Injection 4 mg/cm² | Placebo
Number analyzed (Participants) | 20 | 20 | 22 | 22
percentage of participants | 88.9 | 78.9 | 94.7 | 50.0
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.015, Fisher Exact; Difference from Placebo = 38.9, 95% CI 2-sided [12.6 to 65.2]
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.096, Fisher Exact; Difference from Placebo = 28.9, 95% CI 2-sided [0.4 to 57.5]
Statistical Analysis 3: Comparison: Deoxycholic Acid Injection 4 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.003, Fisher Exact; Difference from Placebo = 44.7, 95% CI 2-sided [20.6 to 68.8]

5. Secondary Outcome: Change From Baseline in Skin Laxity Rating
Description: Skin laxity assessment was based on clinical evaluation and palpation of the submental area on the following scale:
  1 = no laxity; 2 = minimal laxity; 3 = moderate laxity; 4 = very lax. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 4, Week 8, Week 12, Week 16 (4 weeks after last treatment) and Week 24 (12 weeks after last treatment)
Population: Safety/mITT population with available data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Deoxycholic Acid Injection 4 mg/cm² | Placebo
Number analyzed (Participants) | 20 | 20 | 22 | 22
units on a scale
  Week 4 | 0.1 [-0.1 to 0.3] | -0.1 [-0.4 to 0.1] | 0.0 [-0.2 to 0.3] | -0.2 [-0.4 to 0.0]
  Week 8 | 0.1 [-0.1 to 0.4] | -0.1 [-0.4 to 0.1] | 0.1 [-0.1 to 0.3] | -0.1 [-0.4 to 0.1]
  Week 12 | 0.1 [-0.1 to 0.3] | 0.1 [-0.2 to 0.3] | 0.0 [-0.2 to 0.2] | -0.3 [-0.5 to -0.1]
  Week 16 | 0.1 [-0.2 to 0.3] | -0.2 [-0.4 to 0.0] | 0.0 [-0.2 to 0.2] | 0.0 [-0.3 to 0.2]
  Week 24 | 0.1 [-0.2 to 0.3] | -0.3 [-0.5 to 0.0] | 0.0 [-0.2 to 0.2] | -0.1 [-0.4 to 0.1]
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Week 4; Test type: Superiority or Other; p = 0.078, Repeated measures; Based on repeated measures analysis of variance with treatment, visit, center, treatment x visit as fixed effects and subject as a random effect; LS Mean Difference = 0.3, 95% CI 2-sided [0.0 to 0.6]
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Week 4; Test type: Superiority or Other; p = 0.781, Repeated easures; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.4]
Statistical Analysis 3: Comparison: Deoxycholic Acid Injection 4 mg/cm² vs Placebo; Week 4; Test type: Superiority or Other; p = 0.146, Repeated measures; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.1 to 0.5]
Statistical Analysis 4: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Week 8; Test type: Superiority or Other; p = 0.076, Repeated measures; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 0.3, 95% CI 2-sided [0.0 to 0.6]
Statistical Analysis 5: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Week 8; Test type: Superiority or Other; p = 0.975, Repeated measures; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.3]
Statistical Analysis 6: Comparison: Deoxycholic Acid Injection 4 mg/cm² vs Placebo; Week 8; Test type: Superiority or Other; p = 0.183, Repeated measures; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.1 to 0.5]
Statistical Analysis 7: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Week 12; Test type: Superiority or Other; p = 0.017, Repeated measures; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 0.4, 95% CI 2-sided [0.1 to 0.7]
Statistical Analysis 8: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Week 12; Test type: Superiority or Other; p = 0.022, Repeated measures; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 0.4, 95% CI 2-sided [0.1 to 0.7]
Statistical Analysis 9: Comparison: Deoxycholic Acid Injection 4 mg/cm² vs Placebo; Week 12; Test type: Superiority or Other; p = 0.081, Repeated measures; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 0.3, 95% CI 2-sided [0.0 to 0.6]
Statistical Analysis 10: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Week 16; Test type: Superiority or Other; p = 0.510, Repeated measures; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.2 to 0.4]
Statistical Analysis 11: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Week 16; Test type: Superiority or Other; p = 0.330, Repeated measures; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.2]
Statistical Analysis 12: Comparison: Deoxycholic Acid Injection 4 mg/cm² vs Placebo; Week 16; Test type: Superiority or Other; p = 0.720, Repeated Measures; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.4]
Statistical Analysis 13: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Week 24; Test type: Superiority or Other; p = 0.205, Repeated measures; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.1 to 0.5]
Statistical Analysis 14: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Week 24; Test type: Superiority or Other; p = 0.410, Repeated measures; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.5 to 0.2]
Statistical Analysis 15: Comparison: Deoxycholic Acid Injection 4 mg/cm² vs Placebo; Week 24; Test type: Superiority or Other; p = 0.436, Repeated measures; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.2 to 0.4]

6. Secondary Outcome: Change From Baseline in the Cervicomental Angle
Description: The cervicomental angle was measured using a profile view photograph obtained at each visit. A goniometer was used to determine the angle. Cervicomental angle measurements less than 80 degrees are excluded, due to error in measurement.
Time Frame: Baseline and 4 weeks after last treatment (up to 16 weeks after first dose)
Population: Safety/mITT population with available data
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Deoxycholic Acid Injection 4 mg/cm² | Placebo
Number analyzed (Participants) | 7 | 11 | 8 | 13
degrees | -0.7 (3.45) | 2.3 (13.67) | 6.9 (10.67) | -2.3 (9.71)
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection 1 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.762, ANCOVA; Based on analysis of covariance (ANCOVA) model with treatment as fixed effect and baseline SMF rating as covariate; LS Mean Difference = 1.6, 95% CI 2-sided [-9.1 to 12.3]
Statistical Analysis 2: Comparison: Deoxycholic Acid Injection 2 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.248, ANCOVA; Based on analysis of covariance (ANCOVA) model with treatment as fixed effect and baseline SMF rating as covariate; LS mean Difference = 5.2, 95% CI 2-sided [-3.8 to 14.2]
Statistical Analysis 3: Comparison: Deoxycholic Acid Injection 4 mg/cm² vs Placebo; Test type: Superiority or Other; p = 0.061, ANCOVA; Based on analysis of covariance (ANCOVA) model with treatment as fixed effect and baseline SMF rating as covariate; LS Mean Difference = 9.3, 95% CI 2-sided [-0.4 to 19.1]

7. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Values, Weight, Vital Signs, and Physical Examinations
Time Frame: From the first dose of study drug until 12 weeks after the last dose (up to 24 weeks after first treatment).
Population: Safety/mITT population
Measure: Number; unit: participants
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Deoxycholic Acid Injection 4 mg/cm² | Placebo
Number analyzed (Participants) | 20 | 20 | 22 | 22
participants
  Laboratory Values | 0 | 0 | 1 | 0
  Weight | 0 | 0 | 0 | 0
  Vital Signs | 0 | 0 | 0 | 0
  Physical Examinations | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 12 weeks after the last dose (up to 24 weeks after first treatment).
Arm/Group | Deoxycholic Acid Injection 1 mg/cm² | Deoxycholic Acid Injection 2 mg/cm² | Deoxycholic Acid Injection 4 mg/cm² | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 20/20 | 19/20 | 22/22 | 20/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deoxycholic Acid Injection 1 mg/cm² (N=20) | Deoxycholic Acid Injection 2 mg/cm² (N=20) | Deoxycholic Acid Injection 4 mg/cm² (N=22) | Placebo (N=22)
Injection Site Pain (General disorders) | 19 | 16 | 19 | 17
Injection Site Swelling (General disorders) | 17 | 17 | 19 | 10
Injection Site Haematoma (General disorders) | 15 | 15 | 18 | 12
Injection Site Anaesthesia (General disorders) | 17 | 13 | 17 | 4
Injection Site Induration (General disorders) | 8 | 6 | 10 | 2
Injection Site Nodule (General disorders) | 6 | 6 | 7 | 0
Injection Site Erythema (General disorders) | 3 | 5 | 6 | 2
Injection Site Pruritus (General disorders) | 1 | 1 | 3 | 0
Injection Site Paraesthesia (General disorders) | 1 | 1 | 2 | 0
Injection Site Oedema (General disorders) | 2 | 1 | 0 | 1
Injection Site Discomfort (General disorders) | 0 | 1 | 1 | 0
Influenza Like Illness (General disorders) | 1 | 0 | 0 | 0
Injection Site Haemorrhage (General disorders) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 1 | 2 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0
Tonsillitis (Infections and infestations) | 2 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 4 | 3
Migraine (Nervous system disorders) | 1 | 1 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Monoplegia (Nervous system disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Study Agreement requires that the investigator or institution obtain written consent from Kythera prior to presenting and/or publishing results of this study.